CLINICAL TRIAL: NCT03499327
Title: Human Intervention Study to Increase 25-hydroxyvitamin D Levels by Regular Consumption of Wheat Germ Oil (UV-treated) vs. Wheat Germ Oil Untreated (Control)
Brief Title: Human Intervention Study to Increase 25-hydroxyvitamin D Levels
Acronym: WeKo
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Jena (Other)
Collaborators: Martin-Luther-Universität Halle-Wittenberg (Other)
Responsible Party: Principal Investigator, Christine Dawczynski,PhD, Head of the Junior Research Group Nutritional Concepts, University of Jena
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: H5_18
Record Dates: First submitted 2018-03-29; First posted 2018-04-17 (Actual); Last update posted 2023-02-22 (Actual); Status verified 2023-02

CONDITIONS: Vitamin D3 Deficiency
Keywords: vitamin D; ergosterol; 7-dehydro-cholesterol; wheat germ oil
MeSH Terms: interventions — wheat germ oil

STUDY DESIGN:
Intervention Model Description: The randomized, single-blind human intervention study will be conducted in parallel design.
  Half of the participants (n = 17) will consume wheat germ oil UV-treated (intervention) and half of the participants (n = 17) will consume wheat germ oil untreated (placebo). The daily dosage of wheat germ oil is 10 ml and the study products will be consumed over an entire period of 6 weeks (no follow-up).
  The third group (n = 16) do not receive any study products (control).
Who Masked: Participant
Masking Description: The wheat germ oil is dispensed in dark glass bottles without label. The distinction between the groups is based on the expiration date (08.05.2018 vs. 09.05.2018).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Wheat germ oil (UV treated) (Active Comparator): Wheat germ oil (UV treated)
  Interventions: Dietary Supplement: Wheat germ oil (UV treated)
- Wheat germ oil (untreated) (Placebo Comparator): Wheat germ oil (untreated)
  Interventions: Dietary Supplement: Wheat germ oil (untreated)
- Control (No Intervention): no study products

INTERVENTIONS:
Dietary Supplement: Wheat germ oil (UV treated) — Wheat germ oil is naturally rich in vitamin D precursors (ergosterol and 7-dehydrocholesterol), which are converted into vitamin D2 and vitamin D3 by a defined UV light irradiation for the present study (wheat germ oil (UV treated).
  The wheat germ oil (UV treated) is dispensed in dark glass bottles without label. The distinction between the groups is based on the expiration date (08.05.2018 vs. 09.05.2018). The distinction between the groups is not possible for the participants.
  The daily dosage of wheat germ oil is 10 ml and the study products will be consumed over an entire period of 6 weeks (no follow-up).
  Recommendation for intake: pure before a main meal.
  Arms: Wheat germ oil (UV treated)
Dietary Supplement: Wheat germ oil (untreated) — commercial available wheat germ oil The wheat germ oil (untreated) is dispensed in dark glass bottles without label. The distinction between the groups is based on the expiration date (08.05.2018 vs. 09.05.2018). The distinction between the groups is not possible for the participants.
  The daily dosage of wheat germ oil is 10 ml and the study products will be consumed over an entire period of 6 weeks (no follow-up).
  Recommendation for intake: pure before a main meal.
  Arms: Wheat germ oil (untreated)

SUMMARY:
The interventional study will evaluate effectiveness and potential of a regularly consumption of wheat germ oil (UV treated) vs. wheat germ oil (UV untreated) to increase plasma vitamin D levels ín humans.

DETAILED DESCRIPTION:
The interventional study in parallel design will evaluate the effectiveness and potential of a daily consumption of wheat germ oil (UV treated vs. untreated) to increase plasma vitamin D levels in humans.

Wheat germ oil is naturally rich in vitamin D precursors (ergosterol and 7-dehydrocholesterol), which are converted into vitamin D2 and vitamin D3 by a defined UV light irradiation for the present study.

Half of the participants will consume UV-treated wheat germ oil (intervention) and the other part will consume traditional wheat germ oil (untreated, control). The subjects will consume 10 ml of wheat germ oil per day over an entire period of 6 weeks (no follow-up).

On the basis of the planned human intervention study (randomized, single-blind, parallel design) it will be investigated to what extent a regular consumption of wheat germ oil (UV-treated) can contribute to the increase of plasma 25 (OH) D levels.

The comparison is made against the intake of traditional (untreated) wheat germ oil (control).

The study fits with the strategy of the Competence Cluster for Nutrition and Cardiovascular Health (nutriCARD), Halle-Jena-Leipzig, Germany (www.nutriCARD.de) and the study collaborators are active members of the nutriCARD cluster.

ELIGIBILITY:
Inclusion Criteria:

* healthy subjects
* plasma 25(OH) vitamin D < 50 nmol/l
* nutritional habits: western diet

Exclusion Criteria:

* intake of lipid-lowering medications
* gastrointestinal diseases, diabetes mellitus type I and II
* intake of supplements (vitamin D supplements, fish oil capsules, vitamins and minerals) 3 months before and during the study
* relevant food allergies / intolerances
* visit to the solarium (within 4 weeks before beginning of the study and during the study)
* stay in the mountains / skiing (within 4 weeks before beginning of studies and during the study)

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 50 (Actual)
Dates: Start 2018-03-05 (Actual); Primary Completion 2018-04-30 (Actual); Study Completion 2018-04-30 (Actual)

PRIMARY OUTCOMES:
Vitamin D status | change from baseline after 3 and 6 weeks
  plasma levels of 25OHD2, 25OHD3 (nmol/l)

SECONDARY OUTCOMES:
Blood lipids | change from baseline after 3 and 6 weeks
  total cholesterol, LDL cholesterol, HDL cholesterol, triacylglycerides (mmol/L)
Blood glucose | change from baseline after 3 and 6 weeks
  fasting blood glucose (mmol/l)
Insulin | change from baseline after 3 and 6 weeks
  insulin (units/ml)
soluble Klotho (sKlotho) | change from baseline after 3 and 6 weeks
  sKlotho is a component of the FGF23 system and is associated with longevity
Fibroblast growth factor 23 (FGF23) | change from baseline after 3 and 6 weeks
  FGF23 is a regulator of vitamin D metabolism and also a risk factor for heart failure
Fatty acid distribution (erythrocytes) | change from baseline after 3 and 6 weeks
  fatty acid distribution in erythrocyte lipids (% fatty acid methyl ester)
Vitamin D forms 1 | change from baseline after 3 and 6 weeks
  1,25(OH)2D2 (nmol/l)
Vitamin D forms 2 | change from baseline after 3 and 6 weeks
  1,25(OH)2D3 (nmol/l)
Vitamin D forms 3 | change from baseline after 3 and 6 weeks
  24,25(OH)2D (nmol/l)
Vitamin D forms 4 | change from baseline after 3 and 6 weeks
  20(OH)D (nmol/l)

CONTACTS AND LOCATIONS:
Locations (1):
- Friedrich-Schiller-University, Jena, Thuringia, Germany

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Bailer AC, Philipp S, Staudt S, Weidauer T, Kiehntopf M, Lorkowski S, Stangl GI, Dawczynski C. UVB-exposed wheat germ oil increases serum 25-hydroxyvitamin D2 without improving overall vitamin D status: a randomized controlled trial. Eur J Nutr. 2022 Aug;61(5):2571-2583. doi: 10.1007/s00394-022-02827-w. Epub 2022 Feb 27. PMID 35220442
- See also: Study results — https://link.springer.com/article/10.1007/s00394-022-02827-w